CLINICAL TRIAL: NCT06740864
Title: Induction and Stabilization of Gamma Oscillations With 40 Hz Transcranial Alternating Current Stimulation in Healthy Elderly
Brief Title: 40 Hz Transcranial Alternating Current Stimulation for Inducing Gamma Oscillations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Technical University of Dortmund (Other); Leibniz Research Centre for Working Environment and Human Factors (Other); Institute for Research in Fundamental Sciences (IPM) (Unknown)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, Technical University of Dortmund
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IfADo_196_P3
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease; Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 40 Hz prefrontal Transcranial alternating current stimulation (Active Comparator): During prefrontal tACS, an alternating electrical current with a 1 milliamp peak-to-peak amplitude will be delivered, featuring a 15-second ramp-up at the start and a 15-second ramp-down at the end. The stimulation duration is 20 minutes and four channels are used for delivering sinusoidal alternating currents to the head. The alternating current was delivered to the prefrontal cortex bilaterally with the electrodes at F3 and F4 and the return electrodes were placed at the ipsilateral mastoids at TP9 and TP10 (international 10-20 EEG electrode placement system).
  Interventions: Device: Transcranial alternating current stimulation
- 40 Hz frontal-temporal Transcranial alternating current stimulation (Active Comparator): During frontal-temporal tACS, an alternating electrical current with a personalized peak-to-peak stimulation intensity will be delivered, featuring a 15-second ramp-up at the start and a 15-second ramp-down at the end. The stimulation duration is 20 minutes and four channels are used for delivering sinusoidal alternating currents to the head. The alternating current was delivered to the prefrontal and temporal cortices with the active electrodes at AF3-T7 and the return electrodes over AF4-T8 (according international 10-20 EEG electrode placement system).
  Interventions: Device: Transcranial alternating current stimulation
- sham Transcranial alternating current stimulation (Sham Comparator): During sham tACS, an alternating artificial electrical current will be delivered, only ramping the current for 15 seconds up and 15 seconds down at the beginning and end of the stimulation respectively.
  Interventions: Device: Sham Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current will be delivered utilizing a Starstim 8-channel constant current, battery-powered electric stimulator (Neuroelectrics, Barcelona, Spain). Circular carbon rubber electrodes (2cm radius, 12,57 cm2) are used throughout the stimulation.
  Arms: 40 Hz prefrontal Transcranial alternating current stimulation
Device: Transcranial alternating current stimulation — Transcranial alternating current will be delivered utilizing a Starstim 8-channel constant current, battery-powered electric stimulator (Neuroelectrics, Barcelona, Spain). Circular carbon rubber electrodes (2cm radius, 12,57 cm2) are used throughout the stimulation.
  Arms: 40 Hz frontal-temporal Transcranial alternating current stimulation
Device: Sham Transcranial alternating current stimulation — Sham tACS will be applied by only ramping the current for 15 seconds up and 15 seconds down at the beginning and end of the stimulation respectively.
  Arms: sham Transcranial alternating current stimulation

SUMMARY:
This study aims to compare the efficacy of different 40 Hz tACS protocols in entraining gamma oscillations, which are linked to various cognitive functions and play a significant role in cognitive impairments like Alzheimer's disease. Specifically, it examines the effects of 40 Hz tACS applied to frontal brain regions versus fronto-temporal regions on gamma oscillations and working memory in healthy elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* healthy elderly between 50-80 years of age
* normal or corrected to normal eye vision
* right-handed
* non-smokers
* at least 70 % accuracy in working memory training task

Exclusion Criteria:

* history of neurological or psychiatric disorders including seizures or epilepsy,
* Taking CNS, blood pressure and other medications
* having metal implants in the head and neck
* significant cognitive decline meassured by The Montreal Cognitive Assessment (MoCA)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Working Memory behavioral performance | During procedure (20 minutes)
  Participants view a continuous sequence of alphabet letters, presented as stimuli in Arial font, size 120pt, on a tube screen positioned at 60cm eye distance. The stimuli are shown with a time interval of two seconds between them. The task consisted of six blocks with 70 stimuli, including 12 possible hit trials. Participants were instructed to press the left key on a response box if the presented stimulus matched either the one presented one trial prior (1-Back) or three trials prior (3-Back). In all other cases, participants press the right key. The left button is pressed with the index finger, while the right button is pressed with the middle finger of the right hand, with buttons aligned horizontally. The response condition varied by block, with three blocks for 3-Back and three for 1-Back, and the order was counterbalanced across participants and sessions.
electroencephalogram (EEG) oscillatory power | up to 2 hours after the intervention
  Change in the EEG power in the gamma band
electroencephalogram (EEG) functional connectivity | up to 2 hours after the intervention
  Change in EEG functional connectivity, specifically global efficiency, coherence, and phase-locking value at gamma frequency

SECONDARY OUTCOMES:
electroencephalogram (EEG) oscillatory power | up to 2 hours after the intervention
  Change in the EEG power in alpha, delta, theta and beta bands

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Research in Fundamental Sciences, Tehran, Iran